CLINICAL TRIAL: NCT02948049
Title: Accelerometer Based Objective Clinical Outcomes of Spinal Cord Stimulation (SCS) and Peripheral Nerve Stimulation (PNS)
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator resigned from institution
Sponsor: Holy Cross Hospital, Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Actigraph IIT
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Chronic Pain; Back Pain; Neck Pain
Keywords: Accelerometer; Spinal Cord Stimulator; Peripheral Nerve Stimulator; Physical Function
MeSH Terms: conditions — Chronic Pain; Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a single site, prospective, observational trial utilizing a wrist-worn accelerometer to evaluate clinical outcomes of SCS and PNS in the treatment of chronic pain.

DETAILED DESCRIPTION:
Up to 150 evaluable subjects will be recruited at this site on an ongoing basis. Evaluable subjects are defined as subjects that complete the End of Study visit. Each subject will be assigned an accelerometer and have data recorded for a seven-day period pre-implant trial to collect baseline data. The accelerometer will also be worn during the trial for a period of up to seven (7) days. If the trial is successful and the subject is implanted, the subject will wear the accelerometer for a seven-day period at least six (6) weeks post-permanent implant. The following assessments will be administered to subjects at the baseline (pre-implant trial) visit, the end of implant trial visit and the end of study visit (8 weeks post-permanent implant): the Numerical Rating Scale (NRS) 11-point scale for pain; the SF-36 Health Survey; the Oswestry Disability Index (ODI). Subjects treated for neck pain will also complete the Neck Disability Index (NDI). Additionally, the subjects will be asked to complete a subject diary to record average daily NRS scores for days the accelerometer is worn.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study must meet the following criteria:

1. Subject is 18 years of age or older
2. Subject is a candidate for on label use of a SCS or PNS device
3. Subject is ambulatory
4. Subject is able to understand and willing to comply with study procedures and requirements
5. Subject is able to provide informed consent to participate in the study

Exclusion Criteria:

Subjects will be excluded from participation in this study if they meet any one of the following criteria:

1. Subject has comorbidities that, in the judgment of the investigator, may confound the reliability of the information acquired in this study
2. In the judgment of the investigator, the subject is not seeking an improvement in physical function as a treatment goal of SCS or PNS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects recruited for this study will be representative of the population of subjects with chronic pain and a candidate for SCS or PNS trial. Subjects recruited for this study must be 18 years of age or older. It is anticipated that approximately equal numbers of males and females will be recruited. No subjects will be excluded based upon his/her race or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Assess whether there is an increase in objective measurements of physical function in subjects after treatment with an FDA-approved spinal cord stimulation device (SCS) or FDA-approved peripheral nerve stimulation (PNS) device compared with pre-implant. | Pre-implant to 8 weeks post permanent implant
  A subject is considered to have met the primary objective if there is a statistically significant (p value < .05) increase in physical function.

SECONDARY OUTCOMES:
Determine if an increase in physical function obtained from objective assessments of data recorded by the wrist-worn accelerometer in subjects correlate with an improvement in subjective assessments as measured by the Numeric Rating Scale (NRS). | Pre-implant to 8 weeks post permanent implant
Determine if an increase in physical function obtained from objective assessments of data recorded by the wrist-worn accelerometer in subjects correlate with an improvement in subjective assessments as measured by the Short Form-36 Health Survey (SF-36). | Pre-implant to 8 weeks post permanent implant
Determine if an increase in physical function obtained from objective assessments of data recorded by the wrist-worn accelerometer in subjects correlate with an improvement in subjective assessments as measured by the Oswestry Disability Index (ODI). | Pre-implant to 8 weeks post permanent implant
Determine if an increase in physical function obtained from objective assessments of data recorded by the wrist-worn accelerometer in subjects correlate with an improvement in subjective assessments as measured by the Neck Disability Index (NDI). | Pre-implant to 8 weeks post permanent implant

OTHER OUTCOMES:
Evaluate the relationship between physical function and/or pain in subjects stratified into subgroups based on descriptive variables. | Pre-implant to 8 weeks post permanent implant

CONTACTS AND LOCATIONS:
Overall Officials: William P McRoberts, MD, Principal Investigator — Holy Cross Hospital, FL

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Shealy CN, Mortimer JT, Reswick JB. Electrical inhibition of pain by stimulation of the dorsal columns: preliminary clinical report. Anesth Analg. 1967 Jul-Aug;46(4):489-91. No abstract available. PMID 4952225
- [Background] Kumar K, Taylor RS, Jacques L, Eldabe S, Meglio M, Molet J, Thomson S, O'Callaghan J, Eisenberg E, Milbouw G, Buchser E, Fortini G, Richardson J, North RB. The effects of spinal cord stimulation in neuropathic pain are sustained: a 24-month follow-up of the prospective randomized controlled multicenter trial of the effectiveness of spinal cord stimulation. Neurosurgery. 2008 Oct;63(4):762-70; discussion 770. doi: 10.1227/01.NEU.0000325731.46702.D9. PMID 18981888
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Perruchoud C, Buchser E, Johanek LM, Aminian K, Paraschiv-Ionescu A, Taylor RS. Assessment of physical activity of patients with chronic pain. Neuromodulation. 2014 Jun;17 Suppl 1:42-7. doi: 10.1111/ner.12036. PMID 24974774
- [Background] Paraschiv-Ionescu A, Perruchoud C, Buchser E, Aminian K. Barcoding human physical activity to assess chronic pain conditions. PLoS One. 2012;7(2):e32239. doi: 10.1371/journal.pone.0032239. Epub 2012 Feb 23. PMID 22384191
- [Background] Huang KT, Martin J, Marky A, Chagoya G, Hatef J, Hazzard MA, Thomas SM, Lokhnygina Y, Lad SP. A national survey of spinal cord stimulation trial-to-permanent conversion rates. Neuromodulation. 2015 Feb;18(2):133-9; discussion 139-40. doi: 10.1111/ner.12199. Epub 2014 Jun 13. PMID 24930992
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753